CLINICAL TRIAL: NCT04334265
Title: Efficacy and Safety of Anluohuaxian in the Treatment of Rehabilitation Patients With Corona Virus Disease 2019-A Multicenter, Open, Randomized Controlled Study
Brief Title: Efficacy and Safety of Anluohuaxian in the Treatment of Rehabilitation Patients With Corona Virus Disease 2019
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Guiqiang Wang, Principal Investigator, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020 research 110
Record Dates: First submitted 2020-04-01; First posted 2020-04-06 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: Anluohuaxian
MeSH Terms: conditions — COVID-19 | interventions — anluohuaxian

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anluohuaxian combined with regular treatment group (Experimental): Anluohuaxian: 6g each time, twice a day
  Interventions: Drug: Anluohuaxian
- regular treatment group (No Intervention)

INTERVENTIONS:
Drug: Anluohuaxian — 6g each time, twice a day
  Arms: Anluohuaxian combined with regular treatment group

SUMMARY:
To evaluate the efficacy and safety of Anluohuaxian in blocking the progression of pulmonary fibrosis and improving lung function in patients with COVID-19.

DETAILED DESCRIPTION:
In clinical institutions that enroll patients with corona virus disease 2019, two arms, multi-center, randomized and controlled methods are adopted. Patients are divided into two groups, Anluohuaxian combined with regular treatment group and regular treatment group. 750 patients are expected to be enrolled and the cases are allocated according to the ratio of 2( Anluohuaxian combined with regular treatment group): 1(regular treatment group).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed COVID-19, and the nucleic acid test of respiratory specimens such as sputum or nasopharyngeal swabs is negative twice after the treatment (sampling interval is at least 24 hours);
2. Negative nucleic acid test of respiratory specimens such as sputum or nasopharyngeal swabs during screening visits;
3. High-resolution CT of the lung (HRCT) indicates pulmonary fibrosis (thickness of lobular septum, honeycomb-like changes, with or without bronchial / pleural distraction);
4. Voluntarily participate in research and sign informed consent.

Exclusion Criteria:

1. Combined with severe heart, lung (diagnosed with interstitial lung disease, bronchial asthma, chronic obstructive pulmonary disease, etc.), liver and kidney disease or with endocrine, rheumatic, neurologic, malignant and other systemic diseases;
2. Have been diagnosed with connective tissue disease;
3. Pregnant or lactating women;
4. History of mental disorders, substance abuse or dependence;
5. Have used other anti-pulmonary fibrosis drugs in the past 14 days, such as nidanib, pirfenidone, penicillamine, colchicine, tumor necrosis factor alpha blocker, imatinib, glucocorticoid hormones, morphomycodyl esters, azathioprine, cyclophosphamide, interferon-γ, and traditional Chinese medicine;
6. Researchers consider it inappropriate to participate in research;
7. Participating in other clinical research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in high-resolution computer tomography of the lung | 3 months
  Changes in ground-glass shadows, interstitial or air nodules found on high-resolution computer tomography
Change in 6-minute walking distance | 3 months

SECONDARY OUTCOMES:
Changes in compound physiological index | 3 months
Changes in the scores of the St. George's Hospital Respiratory Questionnaire | 3 months
  St. George's Hospital Respiratory Questionnaire range from 0 to 100. 0 stands for no impact on life and 100 stands for extreme impact on life.
Changes in modified British Medical Research Council Dyspnea Scale (mMRC) scores | 3 months
  mMRC score range from 0 to 4. 0 stands for wheezing only when exercising hard and 4 stands for severe breathing difficulties.
Changes in vital capacity of the lung | 3 months
  Adult male vital capacity is about 3,500 ml and female is about 2,500 ml.

CONTACTS AND LOCATIONS:
Overall Officials: Guiqiang Wang, Principal Investigator — Peking University First Hospital
Locations (9):
- China (9):
  - The Second People's Hospital of Fuyang, Fuyang, Anhui
  - Ezhou Central Hospital, Wuhan, Hubei
  - Huoshenshan Hospital of Wuhan, Wuhan, Hubei
  - Jinyintan Hospital of Wuhan, Wuhan, Hubei
  - Tongji Hospital of Huazhong University of Science and Technology, Wuhan, Hubei
  - West Hospital Union Hospital Huazhong University of Science and Technology, Wuhan, Hubei
  - Wuhan Pulmonary Hospital, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Wenzhou Medical University Affiliated First Hospital, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Zhang C, Li J, Wu Z, Wang H, Que C, Zhao H, Wang G. Efficacy and safety of Anluohuaxian in the treatment of patients with severe Coronavirus disease 2019- a multicenter, open label, randomized controlled study: a structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Jun 8;21(1):495. doi: 10.1186/s13063-020-04399-8. PMID 32513299